CLINICAL TRIAL: NCT00963794
Title: Clinical Investigation on a Device for the Diagnosis of Rectal Cancer
Brief Title: Diagnosis of Rectal Cancer by Electromagnetic Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Ermanno Leo, Fondazione IRCCS Istituto Nazionale dei Tumori, Milano
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: INT-D176767
Record Dates: First submitted 2009-08-20; First posted 2009-08-24 (Estimated); Last update posted 2009-08-24 (Estimated); Status verified 2009-08

CONDITIONS: Rectal Cancer
Keywords: Rectal cancer; Population screening; Early detection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electromagnetic measurement (Other): Electromagnetic measurement to detect rectal cancer.
  Interventions: Other: Electromagnetic measurement

INTERVENTIONS:
Other: Electromagnetic measurement — RC screening was carried out using a Tissue Resonance InterferoMeter probe electromagnetic detector, which consists of a nonlinear oscillator placed in a cylindrical probe about 30 cm long, a radiofrequency spectrum analyzer, and dedicated computer software. Detection of RC is based on the decrease of the electromagnetic signal compared to the mean signal obtained in healthy subjects. The test was performed while the patient stood 120 cm from the receiver. The operator was on the opposite side of the examined pelvis. The detector was kept at close contact to the pelvis surface and was moved through six planes, to obtain a scan of the whole pelvis volume. Based on our previous study, we used the electromagnetic detection system at 465 MHz frequency, in a scale from 0 to 255 arbitrary U.
  Other Names: TrimProb

SUMMARY:
The aim of the present prospective study was to evaluate the prediction accuracy of electromagnetic detection of rectal cancer (RC). Eligible subjects were consecutively enrolled in the investigators' Institute and subjected to electromagnetic detection followed by colonoscopy and histopathologic analysis of biopsies. A putative RC carrier status was attributed to subjects showing an electromagnetic signal < 50 units (U).

DETAILED DESCRIPTION:
Eligibility criteria: Gastrointestinal disease or clinical symptoms related to colorectal cancer risk. Exclusion criteria consisted of age younger than 18 years, history of psychiatric illness, and preoperative radiotherapy.

Outcome measures: RC screening was carried out using a Tissue Resonance InterferoMeter probe (TRIMprobe) electromagnetic detector (Galileo Avionica, Turin, Italy), which consists of a nonlinear oscillator placed in a cylindrical probe about 30 cm long, a radiofrequency spectrum analyzer, and dedicated computer software. Detection of RC is based on the decrease of the electromagnetic signal compared to the mean signal obtained in healthy subjects. The test was performed while the patient stood 120 cm from the receiver. The operator was on the opposite side of the examined pelvis. No metallic objects were allowed on the patient and no electronic devices were admitted in the test area. The detector was kept at close contact to the pelvis surface and was moved through six planes, to obtain a scan of the whole pelvis volume. Based on the investigators previous study, we used the electromagnetic detection system at 465 MHz frequency, in a scale from 0 to 255 arbitrary U. The device lets the examination limited to the pelvis and we regarded the rectum cutoff within 15 cm from the anal verge.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal disease or clinical symptoms related to colorectal cancer risk.

Exclusion Criteria:

* Age younger than 18 years, history of psychiatric illness, and preoperative radiotherapy.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 442 (Actual)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Electromagnetic detection system at 465 MHz frequency, in a scale from 0 to 255 arbitrary U. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Nazionale Tumori, Milan, MI, Italy

REFERENCES:
- See also: Fondazione IRCCS Istituto Nazionale Tumori, Milan, Italy — http://www.istitutotumori.mi.it/